CLINICAL TRIAL: NCT02733120
Title: Study on Metabolic Processes and Cognitive Functions in Adults and Adolescents With Autism Spectrum Disorder
Brief Title: Metabolic Processes in Adults and Adolescents With Autism Spectrum Disorder
Acronym: ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0542
Record Dates: First submitted 2016-02-01; First posted 2016-04-11 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy matched controls (Experimental): Study Day: The subject will arrive fasted. A catheter will be inserted in the arm for stable isotope infusion and blood sampling. The hand of the arm used for blood sampling will be placed in a thermostatically controlled warmed box that heats the air. Immediately after a baseline blood sample is taken, an infusion with stable isotopes will be administered by the research nurse. Stable isotopes are given to measure amino acid metabolism. Blood samples will be collected before and/or after infusion. Subjects will be asked to complete a list of questions regarding quality of life, mood and depression, diet.
  Interventions: Other: stable isotope infusion
- Adults with Autism Spectrum Disorder (Experimental): The subject will arrive fasted. A catheter will be inserted in the arm for stable isotope infusion and blood sampling. The hand of the arm used for blood sampling will be placed in a thermostatically controlled warmed box that heats the air. Immediately after a baseline blood sample is taken, an infusion with stable isotopes will be administered by the research nurse. Stable isotopes are given to measure amino acid metabolism. Blood samples will be collected before and/or after infusion. Subjects will be asked to complete a list of questions regarding quality of life, mood and depression, diet.
  Interventions: Other: stable isotope infusion

INTERVENTIONS:
Other: stable isotope infusion — stable isotopes such as 15N2, TRP, 2H3-Leucine, L-[2H3]-3-Methylhistidine, 2H2-Glycine, 2-D-hydroxyproline, 1-13C-ketoisocaproic acid (KIC), L-[Guanido-15N2]-Arginine, L-[ureido-13C-2H2]-Citrulline), L-Glutamine-amide-15N, 1,2-13C2-L-Glutamic acid, 1,2-13C2Taurine, and 13C-Urea is given IV simultaneously

SUMMARY:
The objective of this study is to gain preliminary information and knowledge on metabolic profile in ASD. The benefit of this study will be to expand our insight of the potential relationship in metabolic processes and neuropsychological functions in ASD. For example, based on the obtained data of the study we can determine whether there is a link between the tryptophan pathway and cognitive functions in autism. The project is based on a systematic and multidisciplinary approach using tracers for delineating the mechanism by which the metabolism of amino acids like TRP is involved in affective and cognitive functions in ASD. Using an innovative approach to the evaluation of amino acids has not been used in adults with ASD. In addition, the obtained data of the study holds promise to develop specific markers (metabolic and/or neuropsychological) for guiding the identification those individuals with increased risk of developing mood disturbances or cognitive impairment, and for predicting the therapeutic effect of a specific nutritional interventions in subjects with ASD.

DETAILED DESCRIPTION:
This study investigates the metabolic profile of different amino acids and cognitive functions in adults and adolescents with ASD in comparison with age- and gender-matched healthy young adults. The study involves 1 screening visit of approximately 2 hours and 1 study day of 5 hours

The objective is to explore changes in amino acids (e.g. TRP pathway) in ASD and evaluate the function of TRP in neuropsychological functions by using the technique of stable isotope and our newly developed 'single pulse method' with multiple amino acid and keto-acid isotopes.

The aim of this study is to determine the underlying mechanism by which the metabolism of amino acids such as TRP are involved in mood and cognitive functions in ADS.

ELIGIBILITY:
Inclusion Criteria Healthy:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Age 16 years or older
* Ability to walk, sit down and stand up independently
* Ability to lie in supine or elevated position for 4 hours
* Willingness and ability to comply with the protocol

Inclusion criteria subjects with Autism Spectrum Disorder (ASD):

* Healthy high functioning person diagnosed with autism spectrum disorder
* Age 16 years or older
* Ability to walk, sit down and stand up independently
* Ability to lie in supine or elevated position for 4 hours
* Willingness and ability to comply with the protocol

Exclusion Criteria:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy group)
* Failure to give informed consent
* Established diagnosis of Insulin Dependent Diabetes Mellitus
* Metabolic diseases, including hepatic or renal disorders
* Presence of acute illness or metabolically unstable chronic illness
* Presence of fever within the last 3 days
* Pre-planned surgery of procedures that would interfere with the conduct of the study
* Any other condition according to the PI or study physician that would interfere with proper conduct of the study / safety of the patient
* Current alcohol or drug abuse
* Use of protein or amino acid containing nutritional supplements within 5 days prior to the study days
* Use of long-term oral corticosteroids or short course of oral cortico-steroids 4 weeks preceding first test day
* Body Mass Index of < 18.5 or ≥ 40 kg/m2
* Montreal Cognitive Assessment score of < 20

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Tryptophan turnover | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes

SECONDARY OUTCOMES:
leucine turnover | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
Whole body myofibrillar protein breakdown rate (reflecting muscle protein breakdown) | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
glutathione turnover | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
hydroxyproline breakdown (reflecting collagen breakdown) | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
glutamate turnover | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
taurine turnover | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
urea production | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
Group differences in state of mood as measured by the Hospital Anxiety and Depression Scale (HADS), | 1 day
  a fourteen item self-assessment scale. Seven of the items related to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression.
Group differences in learning and memory as measured by Auditory Verbal Learning Test (AVLT) | 1 day
  Auditory Verbal Learning Test (AVLT): a verbal episodic memory test that evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, retention and recognition of information.
Group differences in learning and memory as measured by Controlled Oral Word Association Test (COWAT), | 1 day
  ontrolled Oral Word Association Test (COWAT): The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonetic verbal fluency. The raw score (total and mean words recorded across the three trials) was reported.
Group differences in learning and memory as measured by Digit Span | 1 day
  recall of numbers in the same order (Digit Forward) and in reverse order (Digit Backward). Measures auditory attention and verbal working memory.
Group differences in overall cognitive abilities as measured by Montreal Cognitive Assessment (MoCA) | 1 day
  assesses several cognitive domains and is used for the screening of mild cognitive impairment. Total scores range from 0-30 with lower scores indicating decreased functioning.
Group differences in attention and executive functions as measured by Trail Making Test (TMT), | 1 day
  In Part A, the examinee is instructed to connect a set of 25 circles with numbers as quickly as possible while maintaining accuracy. In Part B, the examinee is instructed to connect a set of 25 circles, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and mental flexibility. The total time in seconds was reported for each measure.
Group differences in attention and executive functions as measured by Stroop Color-Word Test (SCWT), | 1 day
  a word page with words printed in black ink, a color page with blocks printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The total time in seconds was reported for each trial.
Adolescent/Adult Sensory Profile | 1 day
  a standardized self-questionnaire that generates an individualized profile of sensory processing across four quadrants: low registration, sensation seeking, sensory sensitivity, and sensation avoiding.
Group differences in attention and executive functions as measured by Brief-A | 1 day
  a standardized self-report that captures views of an adult's executive functions or self-regulation in his or her everyday environment.
Group differences in attention and executive functions as measured by PASAT | 1 day
  a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

REFERENCES:
- [Derived] Wierzchowska-McNew RA, Engelen MPKJ, Thaden JJ, Ten Have GAM, Deutz NEP. Obesity- and sex-related metabolism of arginine and nitric oxide in adults. Am J Clin Nutr. 2022 Dec 19;116(6):1610-1620. doi: 10.1093/ajcn/nqac277. PMID 36166849